CLINICAL TRIAL: NCT04599959
Title: COVID-19 Tests: a Systematic Comparison of Viral RNA Test Sample Taking for RT-qPCR, in This Case With a Nasopharyngeal Swab or Saliva Collected With Salivette® Cortisol, to Diagnose SARS-CoV-2 Virus Infection
Brief Title: COVID-19 Tests: Nasopharyngeal Swab vs Saliva Collected With Salivette® Cortisol for Viral RNA Sampling for RT-qPCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0352-2150
Record Dates: First submitted 2020-10-22; First posted 2020-10-23 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Comparison of SARS-CoV-2-RNA detectability in Swab and Salivette samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overall (Swab/Saliva) (Experimental)
  Interventions: Diagnostic Test: Sampling of SARS-CoV-2 RNA from nasopharyngeal swab specimen or saliva collected via Salivette Cortisol

INTERVENTIONS:
Diagnostic Test: Sampling of SARS-CoV-2 RNA from nasopharyngeal swab specimen or saliva collected via Salivette Cortisol — Kylt® for detection/confirmation of SARS-CoV-2 cobas® SARS-CoV-2 (PCR) test TaqPath™ COVID-19 CE-IVD RT-PCR kit

SUMMARY:
The main objective of the tests is to establish saliva collection with Salivette® Cortisol.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed and dated before any samples have been taken.
2. Suspected or confirmed SARS-CoV-2 infection by PCR within the past five days.
3. Male and/or female patients aged 18 years and over.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, México, Mexico

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Moroni-Zentgraf P, Keller C, Eschenfelder CC, Walter Muller H, Sigmund R, Galeana-Cadena D, Marquez-Garcia JE, Moncada-Morales A, Zuniga JA. Salivette(R) Cortisol versus oropharyngeal swabbing for the detection of SARS-CoV-2 infection. Expert Rev Mol Diagn. 2023 Jul-Dec;23(11):1011-1014. doi: 10.1080/14737159.2023.2260308. Epub 2023 Oct 24. PMID 37724431
- See also: Click here to connect to Boehringer Ingelheim Clinical Studies Website — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study compared the viral Ribonucleic acid (RNA) test sample taken for Quantitative reverse transcription polymerase chain reaction (RT-qPCR) via a nasopharyngeal swab versus saliva collected with Salivette® Cortisol in the diagnosing of SARS-CoV-2 virus infection.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Overall: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
  Two samples were taken by medical staff from each participant on the test day, one using a swab (oropharyngeal swab) and the other through saliva collected with Salivette® Cortisol. The collected samples were then shipped and analyzed in Germany.
  Additional up to two samples (swab and/or saliva) were taken for each participant on the test day and analyzed in Mexico.
Period: Overall Study
Arm/Group | Overall
Started | 151
Completed | 151
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
Arm/Group | Overall
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Testing Positive or Negative for SARS-CoV-2 Virus From Swab and Saliva Samples - Processed in Mexico
Description: Number of participants testing positive or negative for SARS-CoV-2 virus from sample collected via swab versus saliva sample collected from Salivette® Cortisol, which samples were processed in Mexico.
Time Frame: At baseline (the test day), up to one day.
Population: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry, and whose samples were processed in Mexico.
Measure: Count of Participants; unit: Participants
Groups:
- Swab - Processed in Mexico: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
  Additional up to two samples (swab and/or saliva) were taken for each participant on the test day and analyzed in Mexico.
  Participants whose swab samples were processed in Mexico and had non-missing results were included in this group.
- Saliva - Processed in Mexico: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
  Additional up to two samples (swab and/or saliva) were taken for each participant on the test day and analyzed in Mexico.
  Participants whose saliva samples collected via Salivette® Cortisol were processed in Mexico and had non-missing results were included in this group.
Arm/Group | Swab - Processed in Mexico | Saliva - Processed in Mexico
Number analyzed (Participants) | 151 | 103
Participants
  Positive | 85 | 13
  Negative | 66 | 89
  Ambiguous | 0 | 1

2. Primary Outcome: Percentage of Participants Testing True Positive or True Negative for SARS-CoV-2 Virus From Swab and Saliva Samples - Processed in Germany
Description: Percentage of participants testing true positive or true negative for SARS-CoV-2 virus from Swab and Saliva samples being processed in Germany was reported. The swab sample was used as the reference. Among participants who were tested positive from swab samples, those who were tested positive from saliva samples were classified as "true positive". Among participants tested negative from swab samples, those who were tested negative from saliva samples were then classified as "true negative".
Time Frame: At baseline (the test day), up to one day.
Population: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry, and had both swab and saliva sample that were processed in Germany.
Measure: Number; unit: Percentage of participants
Groups:
- Swab+Saliva - Processed in Germany: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
  Two samples were taken by medical staff from each participant on the test day, one using a swab (oropharyngeal swab) and the other through saliva collected with Salivette® Cortisol. The collected samples were then shipped and analyzed in Germany.
  Participants with both swab and saliva samples and whose samples were processed in Germany and had non-missing results were included in this group.
Arm/Group | Swab+Saliva - Processed in Germany
Number analyzed (Participants) | 141
Percentage of participants
  True positive (sensitivity): number analyzed (Participants) | 69
  True positive (sensitivity) | 52.2
  True negative (specificity): number analyzed (Participants) | 72
  True negative (specificity) | 100.0

ADVERSE EVENTS:
Time Frame: Up to 1 day.
Description: All eligible participants in this study who had been diagnosed with COVID-19 confirmed by polymerase chain reaction (PCR) test within the past 5 days before study entry.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT04599959/Prot_SAP_000.pdf